CLINICAL TRIAL: NCT07129031
Title: Optimization Strategies for Blood Transfusion Protocols in the Emergency Treatment of Hemorrhagic Shock
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, yin wen, chief physician, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20252202
Record Dates: First submitted 2025-08-09; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hemorrhage; Hemorrhagic Shock; Upper Gastrointestinal Bleeding (UGIB)
Keywords: Hemorrhagic shock; transfusion; low-titer O-group whole blood; group of 1:1:1 component; group of ABO- and Rh-compatible whole blood
MeSH Terms: conditions — Hemorrhage; Shock, Hemorrhagic; Gastrointestinal Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group of 1:1:1 component transfusion (Active Comparator): Following the "Chinese Expert Consensus on Emergency Blood Support Models and Transfusion Strategies for Severely Injured Patients (2024 Edition)", implement the massive transfusion protocol (MTP) by transfusing type-specific blood components in a 1:1:1 ratio (red blood cells : plasma : platelets).
  Interventions: Drug: 1:1:1 component transfusion
- group of ABO- and Rh-compatible whole blood (Active Comparator): Administer type-specific whole-blood transfusion in accordance with the "Chinese Expert Consensus on Emergency Blood Support Models and Transfusion Strategies for Severely Injured Patients (2024 Edition)".
  Interventions: Drug: ABO- and Rh-compatible whole blood
- low-titer O-group whole blood (Experimental): During the emergency phase, administer 4 units of low-titer group O whole blood (anti-A/B IgM antibody titer < 1:64); once the patient's blood type is determined, switch to type-specific whole blood.
  Interventions: Drug: low-titer O-group whole blood

INTERVENTIONS:
Drug: low-titer O-group whole blood — Arm Description: During the emergency phase, administer 4 units of low-titer group O whole blood (anti-A/B IgM antibody titer < 1:64); once the patient's blood type is determined, switch to type-specific whole blood.
  Arms: low-titer O-group whole blood
Drug: 1:1:1 component transfusion — Following the "Chinese Expert Consensus on Emergency Blood Support Models and Transfusion Strategies for Severely Injured Patients (2024 Edition)", implement the massive transfusion protocol (MTP) by transfusing type-specific blood components in a 1:1:1 ratio (red blood cells : plasma : platelets).
  Arms: group of 1:1:1 component transfusion
Drug: ABO- and Rh-compatible whole blood — Administer type-specific whole-blood transfusion in accordance with the "Chinese Expert Consensus on Emergency Blood Support Models and Transfusion Strategies for Severely Injured Patients (2024 Edition)".
  Arms: group of ABO- and Rh-compatible whole blood

SUMMARY:
This single-center, prospective, randomized controlled trial was approved by the institutional ethics committee and overseen by an independent data and safety monitoring board. It enrolled patients with hemorrhagic shock caused by trauma or major gastrointestinal bleeding. Using a random-number-table method, participants were allocated to three groups: (1) Control group: standard massive transfusion protocol (MTP) with transfusing type-specific blood components in a 1:1:1 ratio. (2) Type-specific whole-blood group: following emergency ABO typing and cross-matching, type-specific whole blood was transfused. (3) Low-titer group O whole-blood group: in the emergency phase, 4 units of low-titer group O whole blood (anti-A/B IgM titer < 1:64) were infused; after definitive ABO typing, patients were switched to type-specific whole blood. Clinical data were automatically extracted from the electronic medical record system. Primary endpoints were efficacy (28-day survival), timeliness (transfusion waiting time and time to achieve target mean arterial pressure), cost-effectiveness (total blood consumption and transfusion-related expenses), and safety (transfusion-associated adverse events including TRALI and hemolytic reactions).Statistical analyses included Kaplan-Meier survival curves and Cox proportional-hazards regression, adjusting for confounders such as age and disease severity scores. The advantages and disadvantages of each transfusion strategy were evaluated, and an optimized strategy for emergency blood transfusion in hemorrhagic shock was developed. This strategy was peer-reviewed and refined, culminating in a standardized, multidisciplinary, emergency-transfusion protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemorrhagic shock due to trauma or upper gastrointestinal bleeding who meet emergency transfusion criteria (hemoglobin < 7 g/dL or active bleeding).

Age 10-90 years. Time from onset to hospital admission < 24 hours.

Exclusion Criteria:

* Severe underlying diseases (end-stage organ failure or active malignancy). Known coagulopathy or history of severe transfusion reactions. Refusal to participate or inability to complete follow-up.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
survival rate | 24 hours,30 days

CONTACTS AND LOCATIONS:
Overall Officials: lijunjie li, Study Director — Xijing Hospital; liushanshou liu, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data (IPD) will be shared via a public repository (Dryad Digital Repository) no later than 12 months after the primary results publication.
  Participant-level baseline characteristics
  • Age, sex, body-mass index, Injury Severity Score (ISS), baseline hemoglobin, vital signs on arrival, coagulation parameters (INR, platelet count, fibrinogen), lactate.
  Intervention allocation and delivery data • Randomization group, actual blood products transfused (type, volume, sequence, total units), time from randomization to first transfusion.
  Primary and secondary outcomes (28-day follow-up)
  * Vital status at 28 days (alive/dead), date and cause of death if applicable.
  * Time to achieve mean arterial pressure ≥ 65 mmHg, total blood products and crystalloids within 24 h, incidence and date of TRALI, TACO, acute hemolytic reactions, ICU length of stay, hospital length of stay, total transfusion-related costs.
  Safety events
  • All-grade and grade ≥3 ad
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 2026-January 2028
Access Criteria: 1. The IPD and supporting information will be accessible to the following parties:
  * Principal Investigator (PI) and Study Team: The PI and designated members of the study team, including co-investigators, biostatisticians, and data managers, will have access to the IPD and supporting information for the purpose of conducting the study, analyzing data, and preparing reports.
  * Independent Data and Safety Monitoring Board (DSMB): The DSMB will have access to the IPD and supporting information to monitor the safety and efficacy of the study interventions and to provide recommendations based on interim analyses.
  * Ethics Committees: These committees may request access to the IPD and supporting information to ensure compliance with ethical standards and to review the study protocol and conduct.
  * Sponsor and Sponsor's Representatives: The sponsor of the study and their designated representatives may have access to the IPD and supporting information for oversight and monitoring of the study